CLINICAL TRIAL: NCT01874275
Title: Double-blind, Randomized, Placebo-controlled Study of VECTTOR Treatment for Duchenne Muscular Dystrophy
Brief Title: Duchenne Muscular Dystrophy Clinical Trial
Acronym: DMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alan Neuromedical Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VECTTOR DMD2012
Record Dates: First submitted 2013-06-07; First posted 2013-06-11 (Estimated); Results first posted 2015-03-13 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Duchenne Muscular Dystrophy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- VECTTOR (Experimental): nerve stimulator treatment twice daily for duration of study - 365 days
  Interventions: Device: VECTTOR
- Device - sham (Placebo Comparator): placebo treatment - no electrical stimulation treatment twice daily for duration of study, 180 days - if VECTTOR arm experiencing improvement, subjects in Device-Sham arm will be crossed over into the VECTTOR group and followed for an additional 180 days, for a total study involvement (duration) of 365 days>
  Interventions: Device: VECTTOR

INTERVENTIONS:
Device: VECTTOR — The VT-200, or VECTTOR system, delivers electrical stimulation via electrodes on the acupuncture points of a patient's feet/legs and hands/arms to provide symptomatic relief of chronic intractable pain and/or management of post-surgical pain.
  Once these electrodes are placed, the machine determines the appropriate choice of stimulation by automatically measuring body temperatures through the use of thermistors placed on the fingers during a testing sequence.
  Other Names: electrical nerve stimulator

SUMMARY:
The primary objective of this investigation is to assess the effectiveness of transcutaneous electrical nerve stimulation applied using VECTTOR to reduce the symptoms of Duchenne Muscular Dystrophy and reduce the impact of DMD upon the participants' quality of life.

The primary outcome measures will include:

1. increased muscle strength,
2. increased range of joint motions and
3. improved sleep parameters of ASI, N3 and REM.

DETAILED DESCRIPTION:
Muscle Strength and Joint Range of Motion Testing - All muscle and joint testing was performed at the MedCenter Therapy clinic in Houston, Texas. JTech computerized testing system was utilized including Goniometry, Grip testing, Inclinometry, Muscle Testing and Joint Range of Motion testing occurred on Day 0, 30, 60, 90, 180, and repeated at 12 months to determine muscular strength and joint Range of Motion. JTech computerized testing system was chosen on the basis of reliability and accuracy. At each of the testing intervals, the testing was administered by the same technician with the same equipment to all of the participants. Inter-and intra-tester reliability of the JTech computerized testing system has been the subject of multiple studies. Each of which found high ICCs (>0.93) for both inter- and intra-tester reliability.

All sleep studies were performed at Sleep Diagnostics of Texas in The Woodlands, Texas. Prior to the clinical trial, all of the participants spent two nights in the sleep unit and their sleep study examinations were performed. The second night was used as the Day 0 data. Sleep, breathing, arousals and limb movements were scored manually according to guidelines set forth by the American Academy of Sleep Medicine. The sleep studies were repeated at 6 months and 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have Duchenne Muscular Dystrophy diagnosis as confirmed by licensed physician, wheelchair bound, & age 8 - 20 years old.

Exclusion Criteria:

* Active cancer in the area of application of the treatment, infection, skin infection, pregnancy, thrombophlebitis, pacemaker, amputation of any part of feet or hands, taking steroids. In addition, the participant may not be in any other clinical trial during the time they are in this study.

Ages: 8 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Stelly-Seitz, MD, Principal Investigator — Pediatric Physical Medicine and Rehabilitation Houston, Texas
Locations (1):
- Alan Neuromedical, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- VECTTOR: muscle stimulator treatment twice daily for duration of study - 365 days
  VECTTOR: The VT-200, or VECTTOR system, delivers electrical stimulation via electrodes on the acupuncture points of a patient's feet/legs and hands/arms to provide symptomatic relief of chronic intractable pain and/or management of post-surgical pain.
  Once these electrodes are placed, the machine determines the appropriate choice of stimulation by automatically measuring body temperatures through the use of thermistors placed on the fingers during a testing sequence.
- Device - Sham: placebo treatment - no electrical stimulation treatment twice daily for 180 days followed by active treatment for the duration of study, 365 days
  VECTTOR: The VT-200, or VECTTOR system, delivers electrical stimulation via electrodes on the acupuncture points of a patient's feet/legs and hands/arms to provide symptomatic relief of chronic intractable pain and/or management of post-surgical pain.
  Once these electrodes are placed, the machine determines the appropriate choice of stimulation by automatically measuring body temperatures through the use of thermistors placed on the fingers during a testing sequence.
Period: Overall Study
Arm/Group | VECTTOR | Device - Sham
Started | 4 | 2
Completed | 3 | 2
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- VECTTOR - Active: nerve stimulator treatment twice daily for duration of study - 365 days ...
- Device Sham: placebo treatment - no nerve stimulator treatment twice daily for 180 days of study
- Total: Total of all reporting groups
Arm/Group | VECTTOR - Active | Device Sham | Total
Number analyzed (Participants) | 4 | 2 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 2 | 6
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Range of Motion From Baseline to 180 Days
Description: Range of Motion (ROM) testing (Wireless Tracker System) - All muscle and joint testing was performed using the JTech computerized testing system, including Goniometry, Grip Testing, Inclinometry, Muscle Testing and Joint Range of Motion. Testing occurred at Baseline (Day 0), 30, 60, 90 and 180 days to determine changes in joint Range of Motion. JTech computerized testing system determined the joint range of motion by radio signals from a goniometer measuring movement of the participants' joints. 44 separate tests were performed for Range of Motion for each participant at each time interval. The results from the range of motion tests were averaged the percent change from baseline to 180 days. Efficacy is defined as an increase in range of motion.
Time Frame: Baseline to 180 days
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- VECTTOR: nerve stimulator treatment twice daily for duration of study - assessed at 180 days
- Device - Sham: placebo treatment - no electrical stimulation treatment twice daily for 180 days followed by cross-over with active treatment for the next 180 days
Arm/Group | VECTTOR | Device - Sham
Number analyzed (Participants) | 4 | 2
percentage of change | 67 (44.3) | 33 (49.2)

2. Secondary Outcome: Percent Change in Muscle Strength
Description: Muscle strength testing (Wireless Tracker system) - All muscle strength testing was performed using the JTech computerized testing system, including Goniometry, Grip Testing, Inclinometry, Muscle Testing and Joint Range of Motion. Testing occurred at Baseline (Day 0), 30, 60, 90, and 180 days to determine changes in muscle strength. JTech computerized testing system determined the muscle strength by radio signals from a strain gauge measuring strength of the participant's muscles. 44 separate tests were performed for muscle strength for each participant at each time interval. Efficacy is defined as an increase in the strength measurement (pounds) from Baseline to 180 days.
Time Frame: Baseline to 180 days
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- VECTTOR: nerve stimulator treatment twice daily for duration of study
- Device - Sham: placebo treatment - no electrical stimulation treatment twice daily for 180 days followed by muscle stimulator treatment twice daily for 180 days
Arm/Group | VECTTOR | Device - Sham
Number analyzed (Participants) | 4 | 2
percentage of change | 95 (2.16) | 48 (1.08)

3. Other Pre Specified Outcome: Percent Change in Sleep Quality Arousal Statistics Index (ASI) From Baseline to 180 Days
Description: Sleep / Arousal Statistics Index (ASI) description: Sleep Studies were obtained twice before beginning the study. The second sleep study data was used as baseline. A follow up sleep study was obtained after 6 months (180 days) of Active or Placebo VECTTOR treatment. Sleep, breathing, arousal(s), and limb movements were scored manually according to guidelines of the American Academy of Sleep Medicine. The efficacy of the outcome measure of ASI is demonstrated by a percent improvement between Baseline and 180 days. The ASI is measured by the number of times sleep is interrupted per hour.
Time Frame: Baseline to 180 days
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- VECTTOR: nerve stimulator treatment twice daily for duration of study - 180 days
  VECTTOR: The VT-200, or VECTTOR system, delivers electrical stimulation via electrodes on the acupuncture points of a patient's feet/legs and hands/arms to provide symptomatic relief of chronic intractable pain and/or management of post-surgical pain.
  Once these electrodes are placed, the machine determines the appropriate choice of stimulation by automatically measuring body temperatures through the use of thermistors placed on the fingers during a testing sequence.
- Device - Sham: placebo treatment - no electrical stimulation treatment twice daily for 180 days
  VECTTOR: The VT-200, or VECTTOR system, delivers electrical stimulation via electrodes on the acupuncture points of a patient's feet/legs and hands/arms to provide symptomatic relief of chronic intractable pain and/or management of post-surgical pain.
  Once these electrodes are placed, the machine determines the appropriate choice of stimulation by automatically measuring body temperatures through the use of thermistors placed on the fingers during a testing sequence.
Arm/Group | VECTTOR | Device - Sham
Number analyzed (Participants) | 4 | 2
percentage of change | 38 (1.31) | -53 (1.77)
Statistical Analysis 1: Comparison: VECTTOR vs Device - Sham; Test type: Superiority or Other; p = 0.2413, Mixed Models Analysis

4. Secondary Outcome: Percent Change in Percent Range of Motion From Baseline to 365 Days
Description: Range of Motion (ROM) testing (Wireless Tracker System) - All muscle and joint testing was performed using the JTech computerized testing system, including Goniometry, Grip Testing, Inclinometry, Muscle Testing and Joint Range of Motion. Testing occurred at Baseline (Day 0), 30, 60, 90, 180 and 365 days to determine changes in joint Range of Motion. JTech computerized testing system determined the joint range of motion by radio signals from a goniometer measuring movement of the participants' joints. 44 separate tests were performed for Range of Motion for each participant at each time interval. The results from the range of motion tests were averaged the percent change from baseline to 365 days. Efficacy is defined as an increase in range of motion.
Time Frame: Baseline to 365 days
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- VECTTOR: Range of Motion (ROM) testing (Wireless Tracker System) - All muscle and joint testing was performed using the JTech computerized testing system, including Goniometry, Grip Testing, Inclinometry, Muscle Testing and Joint Range of Motion. Testing occurred at Baseline (Day 0), 30, 60, 90, 180 and 365 days to determine changes in joint Range of Motion. JTech computerized testing system determined the joint range of motion by radio signals from a goniometer measuring movement of the participants' joints. 44 separate tests were performed for Range of Motion for each participant at each time interval. The results from the range of motion tests were averaged the percent change from baseline to 365 days. Efficacy is defined as an increase in range of motion.
Arm/Group | VECTTOR
Number analyzed (Participants) | 4
percentage of change | 59 (45.1)

5. Secondary Outcome: Percent Change in Muscle Strength
Description: Muscle strength testing (Wireless Tracker system) - All muscle strength testing was performed using the JTech computerized testing system, including Goniometry, Grip Testing, Inclinometry, Muscle Testing and Joint Range of Motion. Testing occurred at Baseline (Day 0), 30, 60, 90, 180 and 365 days to determine changes in muscle strength. JTech computerized testing system determined the muscle strength by radio signals from a strain gauge measuring strength of the participant's muscles. 44 separate tests were performed for muscle strength for each participant at each time interval. Efficacy is defined as an increase in the strength measurement (pounds) from Baseline to 365 days.
Time Frame: Baseline to 365 days
Measure: Mean (Standard Deviation); unit: percentage of change
Groups:
- VECTTOR: Muscle strength testing (Wireless Tracker system) - All muscle strength testing was performed using the JTech computerized testing system, including Goniometry, Grip Testing, Inclinometry, Muscle Testing and Joint Range of Motion. Testing occurred at Baseline (Day 0), 30, 60, 90, 180 and 365 days to determine changes in muscle strength. JTech computerized testing system determined the muscle strength by radio signals from a strain gauge measuring strength of the participant's muscles. 44 separate tests were performed for muscle strength for each participant at each time interval. Efficacy is defined as an increase in the strength measurement (pounds) from Baseline to 365 days.
Arm/Group | VECTTOR
Number analyzed (Participants) | 4
percentage of change | 110 (1.93)

6. Other Pre Specified Outcome: Sleep Arousal Statistics Index at 365 Days
Description: Sleep / Arousal Statistics Index (ASI) description: Sleep Studies were obtained twice before beginning the study. The second sleep study data was used as baseline. A follow up sleep study was obtained after 6 months (180 days) of Active or Placebo VECTTOR treatment. Sleep, breathing, arousal(s), and limb movements were scored manually according to guidelines of the American Academy of Sleep Medicine. The efficacy of the outcome measure of ASI is demonstrated by a decrease in the value between Baseline and 180 days. The ASI is measured by the number of times sleep is interrupted per hour. Lower ASI values/numbers indicate improved sleep quality.
Time Frame: Baseline to 365 days
Reporting Status: Not Posted, anticipated posting 2015-03

ADVERSE EVENTS:
Time Frame: 1 year
Description: "0" means the total number of participants in which Serious and Others (Not including Serious) Adverse Events were not collected/assessed.
Groups:
- VECTTOR: nerve stimulator treatment twice daily for duration of study - 365 days ...
Arm/Group | VECTTOR | Device - Sham
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No